CLINICAL TRIAL: NCT02787941
Title: Pharmacist-delivered Multifaceted Intervention to Enhance Medication Adherence Among Post-acute Coronary Syndrome Patients in Vietnam: A Randomised Controlled Trial
Brief Title: Pharmacist-led Intervention to Enhance Medication Adherence in Post-acute Coronary Syndrome Patients in Vietnam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Groningen (Other)
Collaborators: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Katja Taxis, Professor of Pharmacotherapy and Pharmaceutical Care, University of Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PI-MA-ACS-Vietnam
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Acute Coronary Syndrome; Medication Adherence
Keywords: acute coronary syndrome; medication adherence; pharmacist-led interventions; Vietnam
MeSH Terms: conditions — Acute Coronary Syndrome; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive the pharmacist-delivered multifaceted intervention with two counselling sessions in addition to usual care.
  Interventions: Behavioral: Pharmacist-delivered multifaceted intervention
- Control group (No Intervention): The control group will receive usual care without the pharmacist-delivered multifaceted intervention.

INTERVENTIONS:
Behavioral: Pharmacist-delivered multifaceted intervention — First counselling: A pharmacist performs a 30-minute in-person counselling within 1 week before discharge including: (1) assessment and giving advice on basic knowledge of acute coronary syndrome: definition, risk factors, possible cardiac events, and prevention; (2) assessment of past experiences of using medications, encouragement and tailored advice; (3) providing support with pill organiser and drug information leaflet; (4) teaching back and correcting misunderstanding.
  Second counselling: A pharmacist performs a 30-minute telephone counselling within 1 week after discharge including: (1) assessment of general and medication-related issues patients concerning; (2) encouragement and tailored advice; (3) teaching back and correcting misunderstanding.
  Arms: Intervention group

SUMMARY:
Adherence to treatment in post-acute coronary syndrome patients has been found to be poor in several studies. Pharmacists play a significant role in enhancing medication adherence and reducing rates of mortality and re-admission to hospital by performing medication reconciliation and tailoring, and patient education. The purpose of this study is to determine the effect of pharmacist-delivered multifaceted intervention on medication adherence and clinical outcomes of post-acute coronary syndrome patients. The study will be designed as a randomised controlled trial with blinded outcome assessors. The population includes patients who survive during hospitalisation with discharge diagnosis of acute coronary syndrome. Pharmacist-delivered multifaceted intervention consists of two counselling sessions within 1 week before and after hospital discharge including medication reconciliation and tailoring, and support with pill organiser and drug information leaflet. Primary outcome measure is the proportion of patients adherent to medication at 1 month after discharge. Secondary outcome measures are the proportions of patients (1) adherent to medication at 3 months after discharge, (2) readmitted to hospital and (3) dying within 3 months after discharge. The investigators also measure (4) the change in quality of life and (5) beliefs about medicines from baseline at 3 months.

DETAILED DESCRIPTION:
Ischemic heart disease, including acute coronary syndrome, is among the leading causes of death worldwide. Several factors have been shown to attribute to early re-admission to hospital for these conditions including comorbidities, insufficient discharge planning, lack of health literacy, and non-adherence to drug therapy. Adherence to treatment in post-acute coronary syndrome patients has been found to be poor in several studies. Pharmacists play a significant role in enhancing medication adherence and reducing rates of mortality and re-admission to hospital by performing medication reconciliation and tailoring, and patient education. The purpose of this study is to determine the effect of pharmacist-delivered multifaceted intervention on medication adherence and clinical outcomes of post-acute coronary syndrome patients in Vietnam.

The study will be designed as a randomised controlled trial with blinded outcome assessors. Random allocation sequence will be generated using the website randomization.com. The participants will be stratified by age (<65 and 65 years or higher) and sex (male and female), and randomised into two parallel groups in a 1:1 ratio via block technique with random permuted blocks of 2, 4 or 6 patients. Investigators who perform patient recruitment and interventions will be concealed the sequence until the intervention is assigned. One group will receive usual care, called control group, while the parallel group will receive pharmacist-delivered multifaceted intervention in addition to usual care, called intervention group.

Participants will be selected from patients who present to the Cardiology Institute at Ho Chi Minh city, Vietnam. The trial will continue till achievement of sample size and 3-month follow-up thereafter. Estimated duration of recruitment is about 12 months from November, 2015 to November, 2016. The investigators will include patients who survive during hospitalisation with discharge diagnosis of acute coronary syndrome.

The intervention group will receive two counselling sessions in-person and via telephone within 1 week before and after hospital discharge. The interventions will be performed by pharmacists and include medication reconciliation and tailoring, and support with pill organiser and drug information leaflet.

Primary outcome measure is the proportion of patients adherent to medication at 1 month after discharge assessed by the Morisky Medication Adherence Scale - 8 items. Secondary outcome measures are the proportions of patients (1) adherent to medication at 3 months after discharge assessed by the Morisky Medication Adherence Scale - 8 items, (2) readmitted to hospital and (3) dying within 3 months after discharge. The investigators also measure (4) the change in quality of life assessed by the EuroQol EQ-5D-3L and (5) beliefs about medicines assessed by the Beliefs about Medicines Questionnaire (BMQ) from baseline at 3 months.

The process of data collection and management at baseline and during follow-up period is summarised in 9 steps as follows: (1) patient list review; (2) patient recruitment; (3) first data collection at baseline (data from patient interviews); (4) random allocation; (5) first counselling (intervention group only); (6) second data collection at baseline (data from medical records); (7) second counselling (intervention group only); (8) first outcome measurement (at 1 month after discharge); (9) second outcome measurement (at 3 months after discharge).

Analysis will be performed using the intention to treat principle. Reasons for dropouts and proportions for each treatment group will be reported. The investigators will compare the differences in proportions of medication adherence and rates of mortality and hospital readmission between intervention and control groups.

All patients taking part in the trial will be required to provide written informed consent at the time of recruitment. Consent form and the study protocol will be submitted to achieve approval from the Institutional Biomedical Research Ethics Committee of Cardiology Institute at Ho Chi Minh city, Vietnam. The participants will have the right to withdraw at any moment during the study period; their inclusion or exclusion from the study will not affect the usual care provided to them.

ELIGIBILITY:
Inclusion Criteria:

* The investigators include patients who survived during hospitalisation with one of the following diagnoses according to coding of the International Classification of Diseases, 10th revision (ICD-10): unstable angina (I20.0), acute myocardial infarction (I21) or subsequent myocardial infarction (I22)

Exclusion Criteria:

* Have discharge diagnosis not unstable angina (I20.0), acute myocardial infarction (I21) and subsequent myocardial infarction (I22)
* Currently participate in another medication adherence study
* Discharge without prescription
* Unwilling to participate the study
* Unable to communicate in Vietnamese
* Unable to identify their own medications
* No telephone number
* Have cognitive impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients adherent to medication at 1 month after discharge as assessed by the Morisky Medication Adherence Scale - 8 items | 1 month

SECONDARY OUTCOMES:
Proportion of patients adherent to medication at 3 months after discharge as assessed by the Morisky Medication Adherence Scale - 8 items | 3 months
Proportion of patients readmitted to hospital of any cause at 3 months. | 3 months
Proportion of patients dying of any cause at 3 months. | 3 months
Change in quality of life from baseline assessed with EuroQol questionnaire EQ-5D-3L at 3 months. | Baseline and 3 months
Change in beliefs about medicines from baseline assessed with the Beliefs about Medicines Questionnaire (BMQ) at 3 months. | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Katja Taxis, PhD, Principal Investigator — Unit PharmacoTherapy, -Epidemiology & -Economics, Faculty of Mathematics and Natural Sciences, University of Groningen, The Netherlands
Locations (1):
- University of Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nguyen T, Nguyen TH, Nguyen PT, Tran HT, Nguyen NV, Nguyen HQ, Ha BN, Pham TT, Taxis K. Pharmacist-Led Intervention to Enhance Medication Adherence in Patients With Acute Coronary Syndrome in Vietnam: A Randomized Controlled Trial. Front Pharmacol. 2018 Jun 21;9:656. doi: 10.3389/fphar.2018.00656. eCollection 2018. PMID 29977205